CLINICAL TRIAL: NCT03322410
Title: Hydratation Status at Initiation of Peritoneal Dialysis: Study of the Role of Peritoneal Permeability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PA17003
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Fluid Overload; Peritoneal Hyperpermeability; Peritoneal Dialysis; Chronic Kidney Disease
Keywords: Fluid overload; Hydratation statud; Peritoneal hypepermeability; Peritoneal dialysis; Impedancemetry
MeSH Terms: conditions — Edema; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Biological: modified Peritoneal Equilibration test

INTERVENTIONS:
Biological: modified Peritoneal Equilibration test — Peritoneal permeability status determined by modified Peritoneal Equilibration test with complete drainage at 60 minutes as described for Twardowsky
  * " High ": D/P creatinine>0,8; D/D0 glucose<0,25
  * " High average ": 0,65< D/P creatinine <0,8; 0,25< D/D0 glucose <0,38
  * " Low average ": 0,5< D/P creatinine <0,65; 0,39< D/D0 glucose < 0,48
  * " Low " : D/P creatinine<0,5 ; D/D0 glucose>0,49.

SUMMARY:
Bioimpedance is recently known to be a reliable, reproducible and validated technic allowing determination of hydratation status in patients with chronic kidney disease treated with peritoneal dialysis (PD). Overhydratation attested by bioimpedance is strongly associated with cardio-vascular morbidity and mortality in patients with PD. Overhydratation might concern more than half of patients at PD initiation, though the underlying mechanism remains unknown.

High peritoneal permeability (HPP) might concern about a third of patients starting a PD, although only a few datas are published on this condition. HPP at initiation of PD is associated with a decrease in both technical and patient survival and might be responsible of ultrafiltration failure. The underlying mechanisms of HPP at initiation of PD also remains unknown.

To our knowledge, the correlation between hydratation status and peritoneal permeability at initiation of peritoneal dialysis remains unknown. Moreover, there is no datas concerning the cinetic evolution of peritoneal permeability; demographic or biologic factors associated with HPP in days and months following PD start.

The aim of the present study is to correlate hydratation status (attested by bioimpedance) and peritoneal permeability at early start of peritoneal dialysis. Thus, we investigated early cinetic of peritoneal permeability at different time point during the first year of peritoneal dialysis and we analyzed the demographical and biological factors associated with HPP and overhydratation during this period.

This study is a prospective, multicentric cohort study. Fourty patients recruited in a two years' period in five centers of nephrology will be included. Hydratation status will be determined with Fluid Overload measurement by bioimpedance technic thanks to BCM system (Fresenius Medical Care®). Peritoneal permeability will be determined by modified Peritoneal Equilibration Test with complete drainage at sixty minutes. Datas will prospectively be collected, including: weight, blood pressure, diuretic posology, diuresis, PD modality, dialysate prescribed.

ELIGIBILITY:
Inclusion criteria:

* End stage chronic kidney disease
* Ambulatory
* Starting a peritoneal dialysis in one of the participant centers
* Accepting the study protocol
* Age > 18yo

Exclusion criteria:

* Age <18yo
* Protected by the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Hydratation status | Day 7
  Fluid overload (FO) measured with BMC bioimpedance system (Fresenius medical care®)
  * FO < 10th percentile = extracellular dehydration
  * 10th percentile < FO < 90th percentile = extracellular normohydration
  * FO > 90th percentile = extracellular hyperhydration

SECONDARY OUTCOMES:
Peritoneal permeability | Day 7
  Peritoneal permeability status determined by modified Peritoneal Equilibration test with complete drainage at 60 minutes as described for Twardowsky
  * " High ": D/P creatinine>0,8; D/D0 glucose<0,25
  * " High average ": 0,65< D/P creatinine <0,8; 0,25< D/D0 glucose <0,38
  * " Low average ": 0,5< D/P creatinine <0,65; 0,39< D/D0 glucose < 0,48
  * " Low " : D/P creatinine<0,5 ; D/D0 glucose>0,49.
Hydratation status | Day 45
  Fluid overload (FO) measured with BMC bioimpedance system (Fresenius medical care®)
  * FO < 10th percentile = extracellular dehydration
  * 10th percentile < FO < 90th percentile = extracellular normohydration
  * FO > 90th percentile = extracellular hyperhydration
Peritoneal permeability | Day 45
  Peritoneal permeability status determined by modified Peritoneal Equilibration test with complete drainage at 60 minutes as described for Twardowsky
  * " High ": D/P creatinine>0,8; D/D0 glucose<0,25
  * " High average ": 0,65< D/P creatinine <0,8; 0,25< D/D0 glucose <0,38
  * " Low average ": 0,5< D/P creatinine <0,65; 0,39< D/D0 glucose < 0,48
  * " Low " : D/P creatinine<0,5 ; D/D0 glucose>0,49.
Hydratation status | Day 365
  Fluid overload (FO) measured with BMC bioimpedance system (Fresenius medical care®)
  * FO < 10th percentile = extracellular dehydration
  * 10th percentile < FO < 90th percentile = extracellular normohydration
  * FO > 90th percentile = extracellular hyperhydration
Peritoneal permeability | Day 365
  Peritoneal permeability status determined by modified Peritoneal Equilibration test with complete drainage at 60 minutes as described for Twardowsky
  * " High ": D/P creatinine>0,8; D/D0 glucose<0,25
  * " High average ": 0,65< D/P creatinine <0,8; 0,25< D/D0 glucose <0,38
  * " Low average ": 0,5< D/P creatinine <0,65; 0,39< D/D0 glucose < 0,48
  * " Low " : D/P creatinine<0,5 ; D/D0 glucose>0,49.

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

IPD SHARING:
Plan to Share IPD: No